CLINICAL TRIAL: NCT02900326
Title: Effect of a Mindfulness-based Stress Reduction (MBSR) Program Combined With Endurance Exercise Training: a Help to Improve Exercise Capacity and Quality of Life in Breast Cancer
Brief Title: Mindfulness-based Stress Reduction (MBSR) Program Combined With Endurance Exercise Training: a Help in Treatment for Breast Cancer
Acronym: MBSR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5970
Record Dates: First submitted 2015-06-16; First posted 2016-09-14 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Exercise capacity; Mindfulness; Quality of life
MeSH Terms: conditions — Breast Neoplasms | interventions — Mindfulness; Quality of Life; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control patients with no intervention (Placebo Comparator): group without intervention
  Interventions: Other: Vo2max measurements; Genetic: Telomerase activity on a blood sample; Other: Quality of life (questionnaires); Other: Cerebral IRMf
- Endurance training program (8 weeks) group (Experimental): only physical training group
  Interventions: Other: Endurance exercise training; Other: Vo2max measurements; Genetic: Telomerase activity on a blood sample; Other: Quality of life (questionnaires); Other: Cerebral IRMf
- MBSR group (mindfulness-based-stress-reduction) (Experimental): only mental training group (8 weeks)
  Interventions: Other: Mindfulness-based-stress-reduction
- Endurance training program combined with MBSR sessions (Experimental): Endurance training program combined with MBSR sessions, during 8 weeks (mindfulness-based-stress-reduction)
  Interventions: Other: Both interventions together

INTERVENTIONS:
Other: Endurance exercise training — In each group, there will be a comparison of aerobic capacity, quality of life (with questionnaires), functional cerebral measurements (fRMI), and telomerase activity between before and after the 8 weeks program
  Arms: Endurance training program (8 weeks) group
Other: Mindfulness-based-stress-reduction
  Arms: MBSR group (mindfulness-based-stress-reduction)
Other: Both interventions together
  Arms: Endurance training program combined with MBSR sessions
Other: Vo2max measurements
  Arms: Control patients with no intervention; Endurance training program (8 weeks) group
Genetic: Telomerase activity on a blood sample
  Arms: Control patients with no intervention; Endurance training program (8 weeks) group
Other: Quality of life (questionnaires)
  Arms: Control patients with no intervention; Endurance training program (8 weeks) group
Other: Cerebral IRMf
  Arms: Control patients with no intervention; Endurance training program (8 weeks) group

SUMMARY:
Integrative approaches to promote wellness and reduce the distress associated with cancer are considered as essential components of cancer care. In case, exercise training has been shown to produce many positive physiological and psychological benefits. Mindfulness-based stress reduction program shows similar beneficial effects, and especially in emotional distress management. The aim of the study is to examine the cumulative effect of an 8 week-exercise-training program combined with an MBSR program on cardio-respiratory fitness and quality of life in women with breast cancer. These effects are thought to be mediated in part through changes in underlying brain processes, that investigators will be put in light. Through telomerase activity, oxidative stress, mitochondrial respiration and blood cytokine level measurements, investigators could expect to better understand the effect of these combined training in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer
* Having completed the chemotherapy period
* Undergoing radiotherapy and/or hormono therapy

Exclusion Criteria:

* Regular physical activity higher than 4 hours per week.
* Any disease cardiac, respiratory, neurological or articular disease, which counteract the muscular training )

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-05-12 (Actual); Primary Completion 2015-05-12 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Evolution of V02 max between inclusion and 8 weeks | 8 weeks
  effect of physical training associated with mental work on physical abilities of patients

CONTACTS AND LOCATIONS:
Overall Officials: LONSDORFER Evelyne, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Physiologie et EFR/ EA 3072 mitochondrie, stress oxydant et protection musculaire, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sibeoni J, Manolios E, Mathe J, Feka V, Vinez MM, Lonsdorfer-Wolf E, Bloch JG, Bayle F, Meunier JP, Revah-Levy A, Verneuil L. The experience of a program combining two complementary therapies for women with breast cancer: An IPSE qualitative study. PLoS One. 2023 Aug 17;18(8):e0285617. doi: 10.1371/journal.pone.0285617. eCollection 2023. PMID 37590246